CLINICAL TRIAL: NCT05911763
Title: Prospective, Observational , Multicenter Study of Effectiveness of Efanesoctocog Alfa on Long-term Joint Health in Patients With Hemophilia A
Brief Title: A Study to Evaluate Impact of Efanesoctocog Alfa on Long-term Joint Health in Participants With Hemophilia A
Status: Active, not recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS17523; U1111-1281-8840 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-05-12; First posted 2023-06-22 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A (Prophylactic treatment): All participants on efanesoctocog alfa prophylactic treatment fulfilling the overall study inclusion/exclusion criteria. The prophylactic cohort will include the following sub-cohorts:
  Sub-cohort A1 (Joint imaging): Participants with severe hemophilia A and joint imaging by Hemophilia Early Arthropathy Detection with Ultrasound (HEAD-US) or Joint Tissue Activity and Damage Exam (JADE) protocol performed within 6 months of initiating treatment with efanesoctocog alfa or within 3 months after initiating treatment with efanesoctocog alfa available.
  Sub-cohort A2 (Children with no prior joint damage):Participants with severe hemophilia A who have no prior joint damage
  Interventions: Drug: Efanesoctocog Alfa BIVV001
- Cohort B (On-Demand treatment): Participants receiving on-demand treatment with efanesoctocog alfa who fulfil the overall study inclusion/exclusion criteria
  Interventions: Drug: Efanesoctocog Alfa BIVV001

INTERVENTIONS:
Drug: Efanesoctocog Alfa BIVV001 — Given per investigator's discretion
  Other Names: ALTUVIIIO

SUMMARY:
This is a prospective, observational, multi-center longitudinal cohort study to describe the real-world effectiveness, safety and treatment usage of efanesoctocog alfa in patients with hemophilia A treated per standard of care in the US and Japan.

Patients will be enrolled in the study after the introduction of efanesoctocog alfa in the hemophilia treatment landscape in each study country. Decision to initiate treatment with commercially available efanesoctocog alfa will be made by the treating physician independently from the decision to include patients in the study. No study medication is provided. The data related to efanesoctocog alfa effectiveness, safety and usage will be collected prospectively during routine visits (expected annual/semi-annual visits) for up to 5 years following enrollment /treatment initiation.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of hemophilia A
* Patients starting efanesoctocog alfa treatment as per standard of care no more than one month prior to the enrollment date, for either on demand or prophylaxis. Patients starting efanesoctocog alfa treatment for a surgery event may also be enrolled only if the treatment is prescribed at enrollment.
* Physician's decision to treat the patient with efanesoctocog alfa is made prior to and independently of participation in the study.
* Signed and dated informed consent provided by the patient, or by the patient's legally acceptable representative for patients under the legal age before any study-related activities are undertaken. Assent should be obtained for pediatric patients according to local regulations.

Exclusion Criteria:

Diagnosed with other known bleeding disorder

* Participation in an investigational medicinal product trial at enrollment visit, or intake of an Investigational Medicinal Product within 3 months prior to inclusion in this study
* Current diagnosis of a FVIII inhibitor, defined as inhibitor titer ≥0.60 BU/mL

"The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial."

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 200 patients from sites in the US and Japan will be enrolled in the study after the introduction of efanesoctocog alfa in the hemophilia treatment landscape in each of these two countries. To generate data for the broad real-world population of individuals with hemophilia A, eligible patients will include all ages, sexes and hemophilia A severities, whether on prophylactic or on-demand therapy or if efanesoctocog alfa is taken perioperatively.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2028-06-06 (Estimated); Study Completion 2030-09-17 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Annualized joint bleeding rate (AjBR) for treated bleeds | Up to 5 years
  Data will be reported for the effectiveness of efanesoctocog alfa prophylaxis on clinical joint status over 5-years for prophylactic cohort
Change from baseline in Annualized joint bleeding rate (AjBR) for all (treated and untreated) bleeds | Up to 5 years
  Data will be reported for the effectiveness of efanesoctocog alfa prophylaxis on clinical joint status over 5-years for prophylactic cohort
Number of Target joint development, resolution and/or recurrence | Up to 5 years
  Data will be reported for the effectiveness of efanesoctocog alfa prophylaxis on clinical joint status over 5-years for prophylactic coho

SECONDARY OUTCOMES:
Change from baseline in the Hemophilia Joint Health Score (HJHS v2.1) total/domains scores | At 1, 2, 3, 4, 5 years
  HJHS total/domain scores will be reported for prophylactic cohorts (A1 ad A2)
Annual Bleeding Rate (ABR) by type for treated bleeds | At 1, 2, 3, 4, 5 years
  Data will be reported for prophylactic cohorts (A1 and A2)
ABR by type all (treated and untreated) bleeds | At 1, 2, 3, 4, 5 years
  Data will be reported for prophylactic cohorts (A1 and A2)
ABR by location for treated bleeds | At 1, 2, 3, 4, 5 years
  Data will be reported for prophylactic cohorts (A1 and A2)
ABR by location for all (treated and untreated) bleeds | At 1, 2, 3, 4, 5 years
  Data will be reported for prophylactic cohorts (A1 and A2)
ABR for all bleeding episodes (including untreated bleeding episodes) | At 1, 2, 3, 4, 5 years
  Data will be reported for prophylactic cohorts (A1 and A2)
Percentage of patients with zero joint bleeds | At 1, 2, 3, 4, 5 years
  Data will be reported for prophylactic cohorts (A1 and A2)
Annualized factor consumption per participant (IU/kg) assessed by prescription during the follow-up period. | At 1, 2, 3, 4, 5 years
  Data will be reported for prophylactic cohorts (A1 and A2)
Annualized injection frequency per participant (assessed by prescription) during the follow- up period | At 1, 2, 3, 4, 5 years
  Data will be reported for prophylactic cohorts (A1 and A2)
Treatment adherence (%) as judged by the physician during the follow-up period | At 1, 2, 3, 4, 5 years
  Data will be reported for prophylactic cohorts (A1 and A2)
Number of injections of efanesoctocog alfa to treat a bleeding episode. | At 1, 2, 3, 4, 5 years
  Data will be reported for prophylactic cohorts (Sub Cohorts A1 and A2)
Total dose of efanesoctocog alfa to treat a bleeding episode. | At 1, 2, 3, 4, 5 years
  Data will be reported for prophylactic cohorts (Sub Cohorts A1 and A2)
Number of injections of efanesoctocog alfa to treat a bleeding episode | At 1, 2, 3, 4, 5 years
  Data will be reported for On-demand cohort
Total dose of efanesoctocog alfa to treat a bleeding episode | At 1, 2, 3, 4, 5 years
  Data will be reported for On-demand cohort
Percentage of bleeding episodes treated with a single injection of efanesoctocog alfa. | At 1, 2, 3, 4, 5 years
  Data will be reported for On-demand cohort
Occurrence of a change in treatment regimen (on-demand to prophylactic or prophylactic to on-demand) at baseline and follow-up. | At 1, 2, 3, 4, 5 years
  Data will be reported for On-demand cohort
Change from baseline in Hemophilia Early Arthropathy Detection with Ultrasound (HEAD-US) total/domain scores | At 1, 2, 3, 4 and 5 years
  HEAD-US total/domain scores will be reported for joint imaging sub cohort
Change from baseline in Hemophilia Early Arthropathy Detection with Joint Tissue Activity and Damage exam (JADE) musculoskeletal ultrasound (MSKUS) (JADE MSKUS) | At 1, 2, 3, 4 and 5 years
  Data will be reported for consenting participants from the joint imaging sub-cohort
Change from baseline in synovial hypertrophy by change in mm thickness AND/OR HEAD-US synovitis domain, AND/OR by JADE MSKUS synovial hypertrophy +/- power doppler signal | At 6 months, 1, 2, 3, 4 and 5 years
  Data will be reported from the consenting participants from the joint imaging sub-cohort
Occurrence of adverse events (AEs) and serious adverse events (SAEs) | Over 5 year period
  The safety and tolerability of efanesoctocog alfa over 5 years evaluated in all participants
Development of inhibitors (neutralizing antibodies directed against factor FVIII as determined via the Nijmegen modified Bethesda assay. | Over 5 year period
  The safety and tolerability of efanesoctocog alfa over 5 years assessed in all participants
Change from baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) pain intensity 3a questionnaire (adults) | At 3 months, 6 months, 1, 2, 3, 4 and 5 years
  Effectiveness of efanesoctocog alfa assessed per participants' PROs in all participants
Change from baseline in Canadian Hemophilia Outcomes-Kids' Life Assessment Tool (CHO-KLAT) 3.0 (boys ≤18 years old) questionnaire (including Parent Proxy) | At 1, 2, 3, 4 and 5 years
  Effectiveness of efanesoctocog alfa assessed per participants' PROs in all participants
Change from baseline in the occurrence of inpatient and outpatient visits, and length of hospital stay related to hemophilia A | At 1, 2, 3, 4 and 5 years
  Healthcare resource use (HCRU) in efanesoctocog alfa related to hemophilia A over a 5-year period
Hemostatic response/physician reported during peri-operative period for surgery (major, minor) with efanesoctocog alfa. | Over a 5 year period
  Data reported to describe the usage and effectiveness of efanesoctocog alfa during the perioperative period
Number of injections required to maintain hemostasis during perioperative period for surgery (major, minor) | Over 5 year period
  Data reported to describe the usage and effectiveness of efanesoctocog alfa during the perioperative period
Dose per injection required to maintain hemostasis during perioperative period for surgery (major, minor) | Over 5 year period
  Data reported to describe the usage and effectiveness of efanesoctocog alfa during the perioperative period
Total efanesoctocog alfa consumption (IU) during perioperative period for surgery (major, minor) | Over 5 year period
  Data reported to describe the usage and effectiveness of efanesoctocog alfa during the perioperative period
Number of blood component transfusions used during perioperative period for surgery | Over 5 year Period
  Data reported to describe the usage and effectiveness of efanesoctocog alfa during the perioperative period
Type of blood component transfusions used during perioperative period for surgery | Over 5 year period
  Data reported to describe the usage and effectiveness of efanesoctocog alfa during the perioperative period
Estimated blood loss (ml) (intraoperative and post-operative period) for major surgery | Over 5 year period
  Data reported to describe the usage and effectiveness of efanesoctocog alfa during the perioperative period
Number of transfusions required for surgery (intraoperative and post-operative period) | Over 5 year period
  Data reported to describe the usage and effectiveness of efanesoctocog alfa during the perioperative period
Duration of hospitalization (major, minor) | Over 5 years period
  Data reported to describe the usage and effectiveness of efanesoctocog alfa during the perioperative period.
Dose per injection required to maintain hemostasis during perioperative period for surgery (major, minor) | Over a 5 year period
  Data reported to describe the usage and effectiveness of efanesoctocog alfa during the perioperative period for On-demand Cohort

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (28):
- United States (28):
  - Banner MD Anderson Cancer Center- Site Number : 8400008, Gilbert, Arizona
  - Loma Linda University- Site Number : 8400015, Loma Linda, California
  - Orthopedic Institute for Children- Site Number : 8400004, Los Angeles, California
  - The Center for Inherited Blood Disorders- Site Number : 8400001, Orange, California
  - University of Colorado Hemophilia and Thrombosis Center- Site Number : 8400019, Aurora, Colorado
  - William A. Shands Hospital at the University of Florida- Site Number : 8400032, Gainesville, Florida
  - Johns Hopkins All Childrens Hospital - Outpatient Care Center - PIN- Site Number : 8400025, St. Petersburg, Florida
  - Rush University Medical Center -1725 W Harrison St- Site Number : 8400014, Chicago, Illinois
  - The Bleeding and Clotting Disorders Institute- Site Number : 8400005, Peoria, Illinois
  - Indiana Hemophilia and Thrombosis Center- Site Number : 8400013, Indianapolis, Indiana
  - University Of Iowa Hospitals And Clinics- Site Number : 8400026, Iowa City, Iowa
  - ~Massachusetts General Hospital- Site Number : 8400017, Boston, Massachusetts
  - Dana Farber and Boston Children's Hospital- Site Number : 8400031, Boston, Massachusetts
  - University of Michigan Hospital - 1500 E Medical Center Dr- Site Number : 8400023, Ann Arbor, Michigan
  - M Health Fairview- Masonic Cancer Clinic - Clinics- Site Number : 8400010, Minneapolis, Minnesota
  - Mayo Clinic - PPDS- Site Number : 8400035, Rochester, Minnesota
  - Mississippi Center For Advanced Medicine - 7731 Old Canton Rd- Site Number : 8400016, Madison, Mississippi
  - University of Nebraska Medical Center - 985400 Nebraska Medical Center- Site Number : 8400009, Omaha, Nebraska
  - Children's Specialty Center - Las Vegas- Site Number : 8400007, Las Vegas, Nevada
  - Weill Cornell Medicine-New York Presbyterian Hospital- Site Number : 8400021, New York, New York
  - Cincinnati Children's Hospital Medical Center - PIN- Site Number : 8400006, Cincinnati, Ohio
  - Hemophilia Center of Western Pennsylvania- Site Number : 8400012, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center- Site Number : 8400003, Nashville, Tennessee
  - University of Texas Southwestern Medical Center-2001 Inwood Rd- Site Number : 8400020, Dallas, Texas
  - University of Texas Southwestern Medical Center- Site Number : 8400011, Dallas, Texas
  - Gulf States Hemophilia and Thrombophilia Center- Site Number : 8400029, Houston, Texas
  - Washington Institute for Coagulation- Site Number : 8400022, Seattle, Washington
  - Blood Center of Wisconnsin- Site Number : 8400027, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org